CLINICAL TRIAL: NCT06135727
Title: Data Collection for Development of Topcon Health Score
Brief Title: Screening Protocol
Status: Terminated | Type: Observational
Why Stopped: limited access to study population
Sponsor: Topcon Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TPCN-2023-001
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Pathology (glaucoma) arm
  Interventions: Device: Maestro2 OCT
- Normal arm
  Interventions: Device: Maestro2 OCT

INTERVENTIONS:
Device: Maestro2 OCT — 3D Wide (12mmx9mm) OCT scan using the Maestro (Topcon, Japan)

SUMMARY:
The objective of this study is to collect data for the development and validation a screening process using aggregate data.

In this study, data collection will encompass both retrospective and prospective approaches across multiple sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 22 years of age or older on the date of data collection (retrospective) or informed consent (prospective).
* For prospective data collection or missing retrospective data collection, subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent.
* BCVA 20/40 or better (each eye).
* Normal eyes to have normal ocular examination in both eyes
* Normal eyes to have IOP ≤ 21 mmHg in both eyes
* Pathology eyes to have clinical diagnosis of mild or moderate glaucoma in at least one eye

Exclusion Criteria:

* For prospective or missing retrospective data collection, subjects unable to tolerate ophthalmic testing.
* Concomitant diseases known to affect the visual field: history of leukemia, dementia, Parkinson's disease, Alzheimer's disease, stroke, or autoimmune diseases.
* History of intraocular surgery (uncomplicated cataract or glaucoma surgeries are accepted)
* Ocular findings or history of co-morbidities, including, but not limited to: uveitis, non-glaucomatous optic neuropathy, trauma, retinal detachment, vein or artery occlusions, wet age-related macular degeneration, geographic atrophy, proliferative diabetic retinopathy, vitreous hemorrhage, severe cataract, severe non-proliferative diabetic retinopathy. Controlled diabetes and hypertension participants can be included.
* Unreliable VF testing and/or poor-quality OCT scans.
* Poor fixation.
* Pathology eyes with severe glaucoma
* Pathology eyes with glaucoma suspect diagnosis
* Pathology eyes with Ocular Hypertensive diagnosis

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with normal eyes and eyes with moderate or severe glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
RNFL and GCL thickness | 1 day
  Using Maestro2 OCT

CONTACTS AND LOCATIONS:
Overall Officials: Mary Durbin, PhD, Study Chair — Topcon Corporation; Nevin W. El-Nimri, OD, PhD, Principal Investigator — Topcon Corporation
Locations (1):
- Topcon, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No